CLINICAL TRIAL: NCT05935605
Title: Comparison of Noninvasively-Obtained Echocardiographic Doppler Parameters With Simultaneously-Measured Invasive Hemodynamics in Patients Referred for Right Heart Catheterization
Brief Title: Pulmonary Hypertension in Left Heart Disease
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Barry Borlaug, Principal Investigator, Mayo Clinic
Other Study IDs: 17-008263; 1R01HL162828-01A1 (NIH)
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Hypertension; Pulmonary Vascular Disease; Left Heart Disease
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples from the pulmonary artery and systemic artery will be collected at rest & during exercise portion of the cardiac catheterization procedure in EDTA tubes & stored for future discovery-based analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- LHD with no PH: Subjects with Left Heart Disease (LHD) and no Pulmonary Hypertension (PH; mean pulmonary artery (PA) pressure ≤20 mmHg) that are already referred for invasive hemodynamic assessment by right heart catheterization for clinical reasons will undergo transthoracic echocardiography and lung ultrasound.
  Interventions: Diagnostic Test: Transthoracic Echocardiography (TTE); Diagnostic Test: Lung ultrasound
- LHD with isolated PVH: Subjects with Left Heart Disease (LHD) and isolated Pulmonary Venous Hypertension (PVH; mean PA pressure>20 mmHg and PVR<3 WU) that are already referred for invasive hemodynamic assessment by right heart catheterization for clinical reasons will undergo transthoracic echocardiography and lung ultrasound.
  Interventions: Diagnostic Test: Transthoracic Echocardiography (TTE); Diagnostic Test: Lung ultrasound
- LHD with vasoactive PVD: Subjects with Left Heart Disease (LHD) and vasoactive Pulmonary Vascular Disease (PVD; mean PA pressure>20 mmHg and PVR≥3 WU with ≥20% reduction in PVR with inhaled nitric oxide) that are already referred for invasive hemodynamic assessment by right heart catheterization for clinical reasons will undergo transthoracic echocardiography and lung ultrasound.
  Interventions: Diagnostic Test: Transthoracic Echocardiography (TTE); Diagnostic Test: Lung ultrasound
- LHD with fixed PVD: Subjects with Left Heart Disease (LHD) and fixed Pulmonary Vascular Disease (PVD; mean PA pressure>20 mmHg, PVR≥3 WU, and PVR reduction of <20% with inhaled nitric oxide) that are already referred for invasive hemodynamic assessment by right heart catheterization for clinical reasons will undergo transthoracic echocardiography and lung ultrasound.
  Interventions: Diagnostic Test: Transthoracic Echocardiography (TTE); Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiography (TTE) — Transthoracic echocardiography using ultrasound waves will be conducted during the rest and exercise phases of the clinically indicated invasive hemodynamic assessment by right heart catheterization to gather additional measurements of right ventricular function.
Diagnostic Test: Lung ultrasound — A lung ultrasound, which uses sound waves to produce images of the lungs, will be used to assess extravascular lung fluid during the rest and exercise phases of the clinically indicated invasive hemodynamic assessment by right heart catheterization.

SUMMARY:
The goal is to compare patients with and without varying severity of pulmonary vascular disease based upon hemodynamic signatures, echocardiographic measures, and lung ultrasound, in tandem with expired gas metabolic testing and blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the cardiac catheterization laboratory for invasive right heart catheterization for any reason.
* Left Heart Disease, defined as one (or more) of the following:

  * Symptomatic HFpEF, defined by signs and symptoms of HF (dyspnea, fatigue), normal left ventricular (LV) EF (≥50% within 12 months of enrollment), and objective evidence of HF fulfilling at least one of the following criteria: Prior hospitalization for decompensated HF treated with intravenous diuretics; Invasively verified HFpEF defined by pulmonary capillary wedge pressure (PCWP) of ≥15 mmHg at rest and/or ≥25 mmHg during exercise; Clinical diagnosis of HFpEF that does not meet criteria i. or ii. but verified with NTproBNP>300 pg/ml in sinus rhythm or >900 pg/ml in AF; H2FPEF score ≥6 or HFA-PEFF score≥5 according to current guidelines.
  * Symptomatic HFrEF, defined by defined by signs and symptoms of HF (dyspnea, fatigue) and reduced EF (<50%).
  * Symptomatic valvular heart disease (VHD), defined by signs and symptoms of HF (dyspnea, fatigue) in tandem with clinically significant aortic or mitral valve disease (regurgitation and/or stenosis).

Exclusion Criteria:

* Patient inability or unwillingness to undergo noninvasive echocardiography, or if echocardiography would, in the opinion of the investigator, somehow compromise the quality of data acquisition for the clinical case.
* WSPH Group 1 Pulmonary hypertension or PH (Pulmonary arterial hypertension; including congenital heart disease)
* Group 3 PH (Hypoxia/Lung disease-related PH)
* Group 4 PH (Thromboembolic PH)
* Group 5 PH (Miscellaneous)
* Clinically significant parenchymal lung disease, hypoxemia, or lung infection
* Amyloid/infiltrative cardiomyopathy
* Acute Myocarditis
* Acute coronary syndrome or revascularization within 90 days
* Use of PH-specific drugs
* Constrictive pericarditis
* High output heart failure
* HF hospitalization within the preceding 30 days
* Severe or greater aortic (AVA < 1.0 cm2, Mean Gradient > 40 mmHg) or severe mitral (MVA < 1.0 cm) stenosis
* Inability or unwillingness to exercise
* Inadequate echocardiographic imaging windows
* Inability or unwillingness to cooperate with breath holding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected Left Heart Disease (LHD) that are already referred for invasive hemodynamic assessment by right heart catheterization for clinical reasons at Mayo Clinic in Rochester, MN will be identified and approached for participation.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Peak Exercise Cardiac Output | Baseline
  Peak exercise cardiac output (L/min) will be measured using the direct Fick technique during the invasive hemodynamic assessment by right heart catheterization.
Peak Exercise Oxygen Consumption (VO2) | Baseline
  Peak exercise VO2 (ml/kg/min) will be measured using expired gas analysis collected during the invasive hemodynamic assessment by right heart catheterization.

SECONDARY OUTCOMES:
Right Ventricular function assessed by Tricuspid Annular Plane Systolic Excursion (TAPSE) | Baseline
  TAPSE is measured as the displacement (in mm) of the lateral tricuspid annulus toward the apex during systole measured using transthoracic echocardiography during the invasive hemodynamic assessment by right heart catheterization.
Right Ventricular function assessed by tricuspid annular plane systolic excursion (TAPSE)/systolic pulmonary artery pressure (PASP) ratio | Baseline
  TAPSE/PASP ratio (mm/mmHg) will be measured using transthoracic echocardiography during the invasive hemodynamic assessment by right heart catheterization.
Extravascular Lung Fluid Content (B-line score) | Baseline
  Extravascular Lung Fluid Content (B-line score) will be measured using lung ultrasound during the invasive hemodynamic assessment by right heart catheterization.
Peripheral venous pressure | Baseline
  Peripheral venous pressure will be measured through a standard upper extremity peripheral IV line. Peripheral venous pressure (PVP) is reported in millimeters of mercury (mmHg)
Right Arterial Pressure (RA) in the upright position | Baseline
  Right Atrial (RA) pressure will be measured during the invasive hemodynamic assessment by right heart catheterization.
Central pressures (RA, PA, and PCWP) in the upright position | Baseline
  The same pressures that are measured in the supine position will be measured in the upright position in a subset of patients. These measures will be obtained at rest and during exercise (for those receiving this).

CONTACTS AND LOCATIONS:
Overall Officials: Barry Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials